CLINICAL TRIAL: NCT01663363
Title: A Prospective Study to Evaluate the Safety and Effectiveness of Wavefront-Guided LASIK Correction of Myopic Refractive Errors With the iDesign Advanced Wavescan Studio™ System and Star S4IR™ Excimer Laser
Brief Title: Safety and Effectiveness of Wavefront-Guided LASIK Corrections of Myopic Refractive Errors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STAR-110-IDMY
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Results first posted 2015-06-26 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Myopia
Keywords: refractive; LASIK
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- wavefront-guided LASIK (Experimental): LASIK correction of myopic refractive errors. Surgeons will perform wavefront-guided LASIK based upon measurement obtained with the iDesign System.
  Interventions: Device: LASIK correction of myopic refractive errors

INTERVENTIONS:
Device: LASIK correction of myopic refractive errors — Surgeons will perform wavefront-guided LASIK based upon measurement obtained with the iDesign System

SUMMARY:
The purpose of this clinical trial is to demonstrate that wavefront-guided LASIK is safe and effective for the correction of myopic refractive errors.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* Best Spectacle Corrected Visual Acuity (BSCVA) of 20/20 or better
* Uncorrected visual acuity (UCVA) of 20/40 or worse
* Less than 0.75D difference between cycloplegic and manifest refraction sphere.
* Demonstration of refractive stability
* Anticipated post-operative stromal bed thickness of at least 250 microns
* Willing and capable of returning for follow-up examinations for the duration of the study.

Exclusion Criteria:

* Women who are pregnant, breast-feeding, or intend to become pregnant over the course of the study
* Concurrent use of topical or systemic medications that may impair healing
* History of any medical conditions that could affect wound healing
* History of prior intraocular or corneal surgery, active ophthalmic disease, or other ocular abnormality
* Evidence of keratoconus, corneal irregularity, or abnormal topography in the operative eye(s)
* Known sensitivity or inappropriate responsiveness to any of the medications used in the post-operative course

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2012-08; Primary Completion 2014-03 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kendra Hileman, PhD, Study Director — Abbott Medical Optics

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 334 eyes were treated among 170 participants.
Period: Overall Study
Arm/Group | Wavefront-guided LASIK
Started | 170 (334 Eyes were treated among 170 participants)
Completed | 170 (334 Eyes were treated among 170 participants)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The number of participants is 170, but 334 eyes were evaluated among these 170 participants.
Arm/Group | Wavefront-guided LASIK
Number analyzed (Participants) | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 169
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 93
Region of Enrollment [Number; unit: participants]
  United States | 170

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Loss of More Than 2 Lines Best Spectacle Corrected Visual Acuity (BSCVA)
Time Frame: 6 Months
Population: Data from 334 eyes of 170 participants are included for the outcome measure "Percentage of Eyes With Loss of More Than 2 Lines Best Spectacle Corrected Visual Acuity (BSCVA)".
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Wavefront-guided LASIK
Number analyzed (Participants) | 170
Number analyzed (eyes) | 334
percentage of eyes | 0 [NA to NA] — Confidence intervals were not calculated because 0% of eyes lost more than 2 lines of BSCVA.

2. Secondary Outcome: Percentage of Eyes With Uncorrected Visual Acuity (UCVA) of 20/40 or Better
Time Frame: 6 Months
Population: Percentage of eyes with UCVA of 20/40 or better. Target for this outcome measure is greater than 85% achieving UCVA of 20/40 or Better. Data from 334 eyes of 170 participants are included for the outcome measure "Percentage of Eyes With Uncorrected Visual Acuity (UCVA) of 20/40 or Better".
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Wavefront-guided LASIK
Number analyzed (Participants) | 170
Number analyzed (eyes) | 334
percentage of eyes | 98.2 [96.1 to 99.3]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Wavefront-guided LASIK
Serious Adverse Events (participants affected / at risk) | 5/334
Other Adverse Events (participants affected / at risk) | 0/334
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wavefront-guided LASIK (N=334)
Primary open angle glaucoma (Eye disorders) | 2 (2) — Protocol defines primary open angle glaucoma as a serious adverse event.
Transient light sensitivity syndrome (Eye disorders) | 2 (2) — Protocol defines transient light sensitivity syndrome as a serious adverse event
Melting of the flap (Eye disorders) | 1 (1) — Protocol defines melting of the flap as a serious adverse event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreement between the Principal Investigator and the Sponsor (or its agents) restricts the PI's rights to discuss or publish trial results until after the trial is completed and requires prior approval from the sponsor.